CLINICAL TRIAL: NCT04379232
Title: Surgical Activity During the Covid-19 Pandemic: Results for 112 Patients in a French Tertiary Care Center: A Retrospective Observational Cohort Study
Brief Title: Surgical Activity During the Covid-19 Pandemic: Results for 112 Patients in a French Tertiary Care Center
Acronym: SurgiCovid
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2020_001
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Digestive Cancer; Gynaecological Cancer; Head and Neck Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Head and Neck Neoplasms | interventions — Mass Screening; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Screening test for covid ( RT PCR and CT Chest) — Each patient was screened before surgery with RT PCR and CT Chest. Post operatively, if symptoms, patients are tested with RT PCR and CT Chest

SUMMARY:
Background

After the emergence of Covid-19 in China, Hubei Province, the epidemic quickly spread to Europe. France was quickly hit and the Croix-Rousse hospital at the Hospices Civils de Lyon was one of the first French university hospital to receive patients infected with Sars-COV2. The predicted massive influx of patients motivated the cancellation of all elective surgical procedures planned to free hospitalization beds and to free intensive care beds. Nevertheless, patients who had to be canceled had to be properly selected to avoid a life threatening. The retained surgical indications were surgical emergencies, oncologic surgery and organ transplantation.

The objective was to describe the organization of the Croix-Rousse hospital to allow the continuation of these surgical activities while limiting the exposure of patients to the Sars Cov2.

ELIGIBILITY:
Inclusion Criteria:

* surgical management
* > 18 years old

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient operated on during Covid pandemic at Croix-Rousse Hospital, hospices civils de Lyon, Lyon, France
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Symptoms of Covid after surgery | Screening test are performed if the patient becomes symptomatic up to 14 days after surgery. In case of symptoms patients are tested within 24 hours.
  Patients are tested with RT PCR and CT Chest if they declare symptoms after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No